CLINICAL TRIAL: NCT02313935
Title: Effects of Cognitive and/or Physical Exercises Blended by Computer Games in Elderly: The LLM Project Neuroscientific Investigations in Thessaloniki, Greece by the LLM Team at the Aristotle University of Thessaloniki
Brief Title: Cognitive/Physical Computer-Game Blended Training of Elderly: Neuroscientific LLM Studies
Acronym: LLM-AUTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek Alzheimer's Association and Related Disorders (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Project Co-ordinator, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 84171-A
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Mild Cognitive Impairment, So Stated; Mild Dementia; Healthy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- LLM (Experimental): LLM training Participants use the FitForAll exergaming computer platform as the physical training component (PTC); Participants use the language adapted Version of the BrainFitness Program as the cognitive training component (CTC)
  Interventions: Other: LLM
- PTC (Experimental): Physical training only. Participants use the FitForAll exergaming computer platform as the physical training component (PTC).
  Interventions: Other: FFA
- CTC (Experimental): Cognitive training only. Participants use the language adapted Version of the BrainFitness Program as the cognitive training component (CTC)
  Interventions: Other: Brain Fitness
- Passive (No Intervention): Passive Control Participants do not receive an intervention serving as passive controls
- Active (Active Comparator): Active Control Participants receive an alternative cognitive training scheme; software was built on purpose by the AUTH team. The software is called VideoGrade and uses YouTube documentaries.
  Interventions: Other: VideoGrade

INTERVENTIONS:
Other: LLM — LLM training Participants use the FitForAll exergaming computer platform as the physical training component (PTC); Participants use the language adapted Version of the BrainFitness Program as the cognitive training component (CTC)
  Other Names: PTC+CTC
  Arms: LLM
Other: FFA — PTC training Participants use the FitForAll exergaming computer platform as the physical training component (PTC)
  Arms: PTC
Other: Brain Fitness — CTC training Participants use the language adapted Version of the BrainFitness Program as the cognitive training component (CTC)
  Arms: CTC
Other: VideoGrade — Active cognitive training by use of the VideoGrade software by AUTH.
  Arms: Active

SUMMARY:
The study involved Information and Communication Technologies (ICT) and more specifically computer exercises blended with game activities. It was hypothesized that ICT facilitated, game blended cognitive and/or physical exercise improves global cognition when compared to control groups; moreover, these improvements may be manifested by brain activity changes; we explored the impact of potential moderators on combined exercise-induced cognitive benefits, as well as, individual/separate training schemes.

DETAILED DESCRIPTION:
The study was conducted in the Thessaloniki (Greece), in various centers. It was part of the Long Lasting Memories (LLM) project (www.longlastingmemories.eu), which was funded by the European Commission (Information and Communication Technologies Policy Support Program (ICT-PSP) for a three year period (2009-2012). It used a pre-post-test design with the between-participant factor group [intervention(s) vs. passive and/or active control]. Post-test was conducted within 2 weeks after completion of the exercise period. Interventions were carried out in Thessaloniki (Greece) within day care centers, hospitals, senior care centers, a memory outpatient center, local parishes, and at participants' homes.

Centers had to provide 8 exercise weeks, with a frequency of at least 2 physical and 3 cognitive exercise sessions per week, resulting in at least 16 physical and 24 cognitive exercise sessions in total.

A similar trial was registered with Clinical Trial Registration: ClinicalTrials.gov Identifier: NCT02267499

ELIGIBILITY:
Inclusion Criteria:

* no severe cognitive impairment [MMSE ≥ 18]
* fluent language skills
* agreement of a medical doctor
* time commitment to the test and exercise protocol.

Exclusion Criteria:

* concurrent participation in another study
* severe physical or psychological disorders which precluded participation in the intervention (i.e., inability to follow instructions)
* unrecovered neurological disorders such as stroke, traumatic brain injury, unstable medication within the past three months
* severe and uncorrectable vision problems, or hearing aid for less than three months.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
overall cognition | 2 Monhths
  Greek versions of the California Verbal Learning Test [CVLT], the Digit Span Test and the Trail Making Test [TMT] were used to assess cognitive outcomes

SECONDARY OUTCOMES:
physical fitness | 2 months / 6+2 months / 12+2 months
  Physical capacity was measured by means of the Senior Fitness Test
Episodic memory | 2 months / 6+2 months / 12+2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (primary outcome)
working memory | 2 months / 6+2 months / 12+2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (primary outcome)
executive function | 2 months / 6+2 months / 12+2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (primary outcome)
Quality of Life | 2 months / 6+2 months / 12+2 months
  WHOQoL
Instrumental Activities of daily living | 2 months / 6+2 months / 12+2 months
  IADL
Depressive symptoms | 2 months / 6+2 months / 12+2 months
  GDS
Brain function | 2 months
  changes in abnormal brain waves that correlate with mild cognitive decline and dementia as measured by EEG and/or ERPs; changes in resting state networks; localisation of brain region activations/de-activations

REFERENCES:
- [Background] Bamidis PD, Vivas AB, Styliadis C, Frantzidis C, Klados M, Schlee W, Siountas A, Papageorgiou SG. A review of physical and cognitive interventions in aging. Neurosci Biobehav Rev. 2014 Jul;44:206-20. doi: 10.1016/j.neubiorev.2014.03.019. Epub 2014 Apr 4. PMID 24705268
- [Background] Ladas A, Frantzidis C, Bamidis P, Vivas AB. Eye Blink Rate as a biological marker of Mild Cognitive Impairment. Int J Psychophysiol. 2014 Jul;93(1):12-6. doi: 10.1016/j.ijpsycho.2013.07.010. Epub 2013 Aug 1. PMID 23912068
- [Result] Frantzidis CA, Vivas AB, Tsolaki A, Klados MA, Tsolaki M, Bamidis PD. Functional disorganization of small-world brain networks in mild Alzheimer's Disease and amnestic Mild Cognitive Impairment: an EEG study using Relative Wavelet Entropy (RWE). Front Aging Neurosci. 2014 Aug 26;6:224. doi: 10.3389/fnagi.2014.00224. eCollection 2014. PMID 25206333
- [Result] Frantzidis CA, Ladas AK, Vivas AB, Tsolaki M, Bamidis PD. Cognitive and physical training for the elderly: evaluating outcome efficacy by means of neurophysiological synchronization. Int J Psychophysiol. 2014 Jul;93(1):1-11. doi: 10.1016/j.ijpsycho.2014.01.007. Epub 2014 Jan 25. PMID 24472698
- [Derived] Klados MA, Styliadis C, Frantzidis CA, Paraskevopoulos E, Bamidis PD. Beta-Band Functional Connectivity is Reorganized in Mild Cognitive Impairment after Combined Computerized Physical and Cognitive Training. Front Neurosci. 2016 Feb 29;10:55. doi: 10.3389/fnins.2016.00055. eCollection 2016. PMID 26973445
- [Derived] Styliadis C, Kartsidis P, Paraskevopoulos E, Ioannides AA, Bamidis PD. Neuroplastic effects of combined computerized physical and cognitive training in elderly individuals at risk for dementia: an eLORETA controlled study on resting states. Neural Plast. 2015;2015:172192. doi: 10.1155/2015/172192. Epub 2015 Apr 7. PMID 25945260
- See also: The LLM project web site — http://www.longlastingmemories.eu/
- See also: The Greek LLM continuation project/business activity — http://www.llmcare.gr